CLINICAL TRIAL: NCT01908504
Title: F Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) for the Delivery of Adaptive Radiation Therapy
Brief Title: Adaptive Pet Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00033339
Record Dates: First submitted 2013-07-19; First posted 2013-07-25 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2019-05

CONDITIONS: Head and Neck Cancers; Lung and Esophagus Cancers; Anal, Cervix, Vulvar, Vaginal, and Endometrium Cancers
MeSH Terms: conditions — Head and Neck Neoplasms; Esophageal Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET-CT (Other)
  Interventions: Other: PET-CT

INTERVENTIONS:
Other: PET-CT — At radiation planning subjects will have a PET-CT. The CT scan - also called computerized tomography or just CT - combines a series of X-ray views taken from many different angles to produce cross-sectional images of the bones and soft tissues inside the body. A PET is a highly specialized imaging technique that uses short-lived radioactive substances (such as FDG a simple sugar labeled with a radioactive atom) to produce three-dimensional colored images of those substances functioning within the body. These images are called PET scans and the technique is termed PET scanning. PET scanning provides information about the body's chemistry not available through other procedures. Unlike CT or MRI (magnetic resonance imaging), techniques that look at anatomy or body form, PET studies metabolic activity or body function.

SUMMARY:
The purpose of this study is to determine the benefit of using positron emission tomography (PET) in addition to the standard (computed tomography) CT to plan radiation therapy for cancer treatment. The information from the PET-CT may allow the investigators to change the radiation plan or the delivery of the radiation to the tumor/tumor site such as the total dose of radiation or the size of the area to receive further radiation. Presently the use of PET scans to adjust radiation therapy during radiation treatment is not standard of care and is being investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of carcinoma
* Patients with local or regional nodal disease are eligible.
* Zubrod Performance Status 0, 1, or 2.
* Age ≥ 18
* Negative serum pregnancy test for women of child bearing potential
* Patient must sign study-specific informed consent prior to study entry.

Exclusion Criteria:

* No gross disease visible on imaging at the start of radiotherapy
* Contraindication to PET
* Complete response by PET achieved with pre-radiation therapy treatment (surgery or chemotherapy)
* Breast feeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2012-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The number of subjects with benefit from an intra-treatment PET-CT | 3 years
  This benefit lies in the potential to adapt the treatment plan based on an intratreatment PET-CT. This may also be of significant prognostic utility, at an early enough time point to potentially alter treatment accordingly.

SECONDARY OUTCOMES:
Locoregional control. | Day of intra treatment PET-CT/ approx 2-4 hours
  This study will evaluate the prognostic value of intra-treatment functional imaging on clinical relevant tumor endpoints (i.e. locoregional control, freedom from distant metastases, and overall survival).Comparison of intra-treatment FDG-PET indices will identify two groups of responses: PET responses and PET non-responses, which will correlate with prognosis.
Freedom from distant metastases | 3 years
  Subjects will be evaluated in regular follow up with repeat imaging as per the standard of care, or at the treating investigator's discretion. Frequency of follow up will be determined by the standard practice for the disease site and stage.
Measure overall survival (OS) | 3 years
  Subjects will be evaluated in regular follow up with the investigators according to the standard of care for each disease site.
Measure acute toxicities | During radiation therapy and within 30 days of the last radiation treatment
  Acute toxicity will be assessed weekly as per the standard practice of the treating investigator.
Measure late toxicities | 3 years
  Subjects will be evaluated in regular follow up with measures of treatment related side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Junzo Chino, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Mowery YM, Vergalasova I, Rushing CN, Choudhury KR, Niedzwiecki D, Wu Q, Yoo DS, Das S, Wong TZ, Brizel DM. Early 18F-FDG-PET Response During Radiation Therapy for HPV-Related Oropharyngeal Cancer May Predict Disease Recurrence. Int J Radiat Oncol Biol Phys. 2020 Nov 15;108(4):969-976. doi: 10.1016/j.ijrobp.2020.08.029. Epub 2020 Aug 13. PMID 32800802